CLINICAL TRIAL: NCT07134348
Title: Evaluation of Sequelae in Permanent Successors Following Traumatic Injuries to Primary Teeth
Status: Completed | Type: Observational
Sponsor: Zeynep Aslı GÜÇLÜ (Other)
Responsible Party: Sponsor-Investigator, Zeynep Aslı GÜÇLÜ, Assoc. Prof., TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: 2024/267
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Dental Trauma; Enamel Hypoplasia; Sequelae; Sequelae Successors
Keywords: deciduous teeth, dental trauma, enamel hypoplasia, sequelae, successors
MeSH Terms: conditions — Dental Enamel Hypoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trauma Group: Children with primary teeth trauma history
- Control Group: no history random observation in clinic.

SUMMARY:
Retrospective data analysis of children with primary dental trauma and follow-up visual examination to find out the sequelae.

DETAILED DESCRIPTION:
An observational study of permanent teeth that have enamel defects, coloration, or developmental disruption after primary tooth injury. A control group without history of trauma or dental injury to compare the enamel defect statistics.

ELIGIBILITY:
Inclusion Criteria:

* • Children who had experienced TDI-p

  * Presence of a permanent tooth germ below the primary teeth
  * Children aged between 5 and 12 years, regardless of sex
  * Patients and their guardians who agreed to participate in follow-up sessions
  * Permanent teeth that had fully erupted according to Von Arx's [16] classification.

Exclusion Criteria:

* • Children with long-term antibiotic use due to chronic illnesses that could cause enamel hypoplasia

  * Children with congenital absence of permanent tooth germs
  * Permanent teeth with caries or restorations due to trauma or other causes
  * Permanent teeth that had not yet erupted or had only partially erupted
  * Children with primary tooth trauma who were unable to attend the follow-up session
  * Children with a history of trauma to their permanent teeth
  * Children without any history of trauma to primary teeth

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Data from 275 traumatized primary teeth of 137 children
  * 101 children were included in the study 36 children excluded because the corresponding permanent successors had not yet erupted, and four permanent teeth and secondary trauma
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
enamel hypoplasia | 2018 and 2022
  developmental enamel defect with color change

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No